CLINICAL TRIAL: NCT02769975
Title: Evaluation of Children With Endocrine and Metabolic-Related Conditions
Status: Recruiting | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 160113; 16-CH-0113
Record Dates: First submitted 2016-05-11; First posted 2016-05-12 (Estimated); Last update posted 2025-09-24 (Actual); Status verified 2025-09-18

CONDITIONS: Adrenal Insufficiency; Growth Disorder; Endocrine Diseases; Metabolic Disease; Bone Diseases, Metabolic
Keywords: Endocrinology; Obesity; Pediatric; Growth Disorder; Pubertal Development
MeSH Terms: conditions — Adrenal Insufficiency; Growth Disorders; Endocrine System Diseases; Metabolic Diseases; Bone Diseases, Metabolic; Obesity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Case Only: Children ages 3 months to 100 with known or suspected endocrine or metabolism disorders. Family members ages 3 months to 100. They may participate in the DNA part of the study

SUMMARY:
Background:

Endocrine glands give off hormones. Researchers want to learn more about the disorders that affect these glands in children. These disorders might be caused by changes in genes. Genes contain DNA, which is the blueprint of how a cell works. Researchers want to identify the genes involved in endocrine and metabolic disorders. This might help develop new ways to diagnose and treat the disorders.

Objective:

To study the inheritance of endocrine or metabolism disorders.

Eligibility:

Children ages 3month-18 with known or suspected endocrine or metabolism disorders.

Family members ages 3months-100. They may participate in the DNA part of the study.

Design:

Participants will be screened with a review of their medical records. Their parents or guardians will allow the records to be released.

Participants will have a clinic visit. This may include a physical exam and medical history.

Parents or guardians will give their consent for the study. Participants may have tests, surgery, or other procedures to help diagnose or treat their condition. These could include:

Blood, urine, and saliva tests

Growth hormone test

Pituitary and adrenal function tests

Picture of chromosomes

Imaging tests. These may include X-ray, ultrasound, scans, or a skeletal survey.

Genetic tests

Sleep study

Medical photographs

If surgery is done, a tissue sample will be taken.

Participants may have follow-up visits for diagnosis and treatment.

Participating relatives will have one visit. This will include medical history and blood and saliva tests. The blood and saliva will be used for DNA testing.

DETAILED DESCRIPTION:
Study Description:

This protocol is designed to allow endocrine-related evaluations of children with known or suspected endocrine or metabolic disorders.

Children with endocrine or metabolic-related condition(s) who may or may not be eligible for a specific NICHD research protocol, may be evaluated under the auspices of this protocol. Standard clinically indicated laboratory or radiological studies may be performed to confirm a diagnosis or to aid in the management of the patient. In some cases, the child participant may receive medical or surgical treatment for their disorder at the National Institutes of Health (NIH) Clinical Center (CC) according to current clinical practice. Family members of children evaluated on this protocol (who have informative meiotic inheritance relationships to the proband or index case) may be enrolled in the genetic/DNA testing part of the protocol.

Objectives:

Primary Objective:

-Comprehensive evaluation of pediatric endocrine diseases and conditions as well as track natural progress of the development of such

conditions in diverse population of pediatric subjects with a known or suspected endocrine or metabolic disorder.

Secondary Objective:

-Samples for molecular genetic or WES testing

Endpoints:

Primary Endpoint:

Appraisal of number and diversity of endocrine related diagnosis of patients evaluated on this protocol.

Secondary Endpoints:

-Number of samples for molecular genetic or WES testing.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* Participants with known or suspected endocrine disorder age 3 months-18 years are eligible for this protocol.
* Relatives ages 3 months-100 years may be enrolled if clinically indicated for the diagnosis of a proband.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Lack of suspected endocrine disorders.
* Any medical, physical, psychiatric, or social conditions, which, in the opinion of the investigators, would make participation in this protocol not in the best interest of the patient, will exclude participation. Patients who are critically ill, unstable, or with severe organ failure that may affect/limit the endocrine evaluation and place unsustainable demands on Clinical Center or NICHD resources will be excluded.

Ages: 3 Months to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children with endocrine or metabolic-related condition(s) who may or may not be eligible for a specific NICHD research protocol, may be evaluated under the auspices of this protocol to advance the clinical skills of physicians participating in NICHD clinical research and training programs, and to provide stimuli for new clinical research initiatives.
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2016-07-12 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Provide an option for patients with unusual or challenging endocrine or metabolic conditions, who may or may not be eligible for an existing research protocol, to be evaluated at NIH. | Baseline
  Provide an option for patients with unusual or challenging endocrine or metabolic conditions, who may or may not be eligible for an existing research protocol, to be evaluated at NIH.
Recruit a diverse population of pediatric subjects with a known or suspected endocrine or metabolic disorder in order to provide NICHD investigators and trainees with hands-on experience related to the diagnosis, management, treatment, and follo... | Baseline
  Recruit a diverse population of pediatric subjects with a known or suspected endocrine or metabolic disorder in order to provide NICHD investigators and trainees with hands-on experience related to the diagnosis, management, treatment, and follow-up of p

SECONDARY OUTCOMES:
All studies or procedures (other than biospecimens/DNA) that are not clinically indicated need to be explicitly described in the protocol or approved by amendment. | Ongoing
  All studies or procedures (other than biospecimens/DNA) that are not clinically indicated need to be explicitly described in the protocol or approved by amendment.
Any prospective (including pilot investigations) or retrospective hypothesis driven research for patients enrolled in this protocol must be approved by the NICHD Office of the Clinical Director and NICHD IRB. | Ongoing
  Any prospective (including pilot investigations) or retrospective hypothesis driven research for patients enrolled in this protocol must be approved by the NICHD Office of the Clinical Director and NICHD IRB.
Clinical evaluation of children with unusual or challenging endocrine or metabolic conditions may include whole exome sequencing (WES) or other new molecular technologies to identify the molecular genetic etiology | Ongoing
  Clinical evaluation of children with unusual or challenging endocrine or metabolic conditions may include whole exome sequencing (WES) or other new molecular technologies to identify the molecular genetic etiology

CONTACTS AND LOCATIONS:
Overall Officials: Catherine M Gordon, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
The protocol does not address an IPD plan.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2016-CH-0113.html